CLINICAL TRIAL: NCT02971826
Title: Use of the Thrombectomy Device ReVive™ SE in the Acute Treatment of Stroke
Acronym: REVIVE SE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL16_0571; 2016-A01470-51 (Other: ID-RCB)
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Stroke; thrombectomy; REVIVETM SE; MRI; Computed Tomography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thrombectomy using the REVIVETM SE device (Experimental): Thrombectomy using the REVIVETM SE device in patient with an ischemic stroke
  Interventions: Device: REVIVETM SE thrombectomy

INTERVENTIONS:
Device: REVIVETM SE thrombectomy — Mechanical thrombectomy using the REVIVETM SE device in patient with an ischemic stroke due to an intracranial arterial occlusion

SUMMARY:
The last marketed thrombectomy devices, named stentretriever, permit a better and faster recanalization in patient with a stroke. The REVIVETM SE is a device designed to restore the brain perfusion in patient with an intracranial artery occlusion. The REVIVETM Se device is not widely use in Europe and in France. The objective of this study is to assess the interest of using this device in the standard care of ischemic stroke in the radiology unit of the hospital Pierre Wertheimer, Lyon. The medical care will not be modified but data will be collected in order to determine whether or not this device is useful for the practice of the radiology unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an ischemic stroke detected by Computed Tomography (CT) or Magnetic Resonance Image (MRI)
* Large proximal arterial occlusion : M1 segment of the Middle cerebral artery (MCA), Internal Carotid Artery (ICA) or Basilar Artery (BA)
* Last known well (without neurological symptoms) ≤ 8 hours of treatment initiation
* Score NIHSS ≥4
* Eligibility on an endovascular procedure using REVIVETM SE device
* No opposition of the patient to participate at the study

Exclusion Criteria:

* Diagnostic cerebral imaging impossible
* Distal occlusion
* Tortuous vessel or other specificity preventing the access of device
* Vessel diameter < 1.5 mm
* Known hypersensibility or allergy to nitinol
* Subjects not covered by or having the right to social security
* Deprivation of civil rights (guardianship, safeguard justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
number of patients with a TICI score of 2b or 3 just after the thrombectomy | up to 2 days
  The TICI score is a grading system which evaluate the degree of reperfusion as seen on arteriography

SECONDARY OUTCOMES:
Number of the other devices use during the thrombectomy (Gidewire, catheter, etc.) | up to 2 days
  Review of the medical report which collected the devices used
Number of other procedures to treat the patient (thrombolysis, thromboaspiration, etc) | Day 0
  Review of the medical report which collected the acute treatments
Time to obtain the appropriate recanalization (TICI 2b or 3) | At the end of the procedure - Day 0
  Time of recanalization reported by the investigator on the medical report

CONTACTS AND LOCATIONS:
Overall Officials: Françis TURJMAN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Neuroradiology unit, Bron, France

IPD SHARING:
Plan to Share IPD: No